CLINICAL TRIAL: NCT01510483
Title: Clinician Promotion of Healthy Diet and Activity to Reduce Obesity Among Adolescents
Brief Title: Clinician Promotion of Healthy Diet and Activity to Reduce Obesity Among Adolescents: HEALTHY SMILES
Acronym: HS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Responsible Party: Principal Investigator, Melbourne Hovell, Director of CBEACH, Distinguished Professor of Public Health, San Diego State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 5R01CA138192 (NIH)
Record Dates: First submitted 2011-11-14; First posted 2012-01-16 (Estimated); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Obesity
Keywords: obesity prevention; tobacco prevention; nutrition; physical activity; sedentary activity; tobacco use; tobacco exposure; prevention; clinician intervention; preteen; adolescents
MeSH Terms: conditions — Obesity; Motor Activity; Tobacco Use

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Obesity prevention (Experimental): Orthodontist promotion of physical activity and healthy diet
  Interventions: Behavioral: Obesity Prevention
- Tobacco prevention (Active Comparator): Orthodontist promotion of tobacco and second hand smoke avoidance
  Interventions: Behavioral: Tobacco Prevention

INTERVENTIONS:
Behavioral: Obesity Prevention — Those in the experimental, obesity prevention, condition will be exposed to the office-wide intervention for diet and activity. The intervention will consist of training of orthodontists and office staff to provide appropriate social prompts, reinforcement and counseling, and modification of the offices to provide supportive physical and social resources for their patients and parents.
  Arms: Obesity prevention
Behavioral: Tobacco Prevention — Those in the control, tobacco prevention, condition will be exposed to the office-wide intervention for avoidance of tobacco and second hand smoke. The intervention will consist of training of orthodontists and office staff to provide appropriate social prompts, reinforcement and counseling, and modification of the offices to provide supportive physical and social resources for their patients and parents.
  Arms: Tobacco prevention

SUMMARY:
This study will test an 18-month intervention designed to increase physical activity, reduce sedentary practices and promote healthy diets or reduce tobacco use and exposure among preteens who obtain orthodontic care. Relevance: If successful, this study may inform policies that would promote all specialists (orthodontists, physicians, general dentists) to deliver brief counseling for diet, physical activity, and tobacco prevention.

DETAILED DESCRIPTION:
This study will test a 18-month multi-component intervention designed to increase physical activity, reduce sedentary practices and promote healthy diets among preteens who obtain orthodontic care. The intervention is based on the Behavioral Ecological Model (BEM), where interacting physiological, environmental, and cultural contingencies select behavior. This study will require five years to recruit 40 orthodontist offices, and 1700 youth, and implement an office-wide intervention for promoting healthy diet and physical activity among 8-14 yr old youth. Our primary aims are to detect a differential change in diet, physical activity and BMI in our experimental group compared to the tobacco prevention control group; to observe differential effects of the intervention between low vs. high SES; and similarly for males vs. females; to validate our primary outcome variables by contrasting them with a "gold standard"; and determine the degree to which family and peer encouragement for sedentary and high caloric diet at baseline increases the relative effect of the orthodontist intervention. Offices will be assigned at random to condition producing a 2 (experimental group) by 2 strata (low vs. high SES) by 2 strata (male vs. female) by 4 (repeated measures) experimental design. Those in the experimental condition will be exposed to the office-wide intervention for diet and activity; those in the control condition will be exposed to an office-wide intervention for tobacco prevention. The intervention will consist of training of orthodontists and office staff to provide appropriate social prompts, reinforcement and counseling, and modification of the offices to provide supportive physical and social resources for their patients and parents. Measures of diet, physical activity, body composition, tobacco use, fitness and family and peer encouragement will occur at baseline, 12, 18, and 24 months. Differential change over time will be analyzed using Random Effects Multivariate modeling. Analyses will include control for office cluster effects and multivariate models will include analyses of hypothetical main effects, experimental group by time interactions, and moderating effects by inclusion of interaction terms for susceptibility by experimental condition and other possible moderators. Relevance: If successful, this study may inform policies that would promote all specialists (physicians, general dentists) to deliver brief counseling for diet and physical activity. Doing so might yield the cumulative exposure necessary to effect and sustain change in a large proportion of the preteen population.

ELIGIBILITY:
Inclusion Criteria:

* 8-14 years old
* receiving orthodontic care at a participating orthodontic office
* at least 1 year left in braces

Exclusion Criteria:

* participating in 9 or more months of structured
* organized sports for 3 or more days a week, youth who have serious conditions that preclude physical activity or make the child incapable of managing his/her own care will not qualify for this study
* individuals who report anorexia, bulimia or severe, diagnosed depression will not be eligible

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 693 (Actual)
Dates: Start 2010-01; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Change in Body Mass Index | Baseline, 2, 4, 6, 8, 10, 12, 14, 16, 18, 24 months
  Body Mass Index assessed at Baseline, 12 month, 18 months and 24 months; and every 6-8 weeks during intervention period.

SECONDARY OUTCOMES:
Change in physical and sedentary activity | Baseline, 12, 18 and 24 months
Change in dietary intake | Baseline, 12, 18 and 24 months
Change in tobacco use and exposure | Baseline, 12, 18 and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Melbourne F Hovell, PhD, MPH, Principal Investigator — SDSU/GSPH
Locations (1):
- SDSU-Center for Behavioral Epidemiology & Community Health, San Diego, California, United States

REFERENCES:
- [Background] Hovell MF, Slymen DJ, Keating KJ, Jones JA, Burkham-Kreitner S, Hofstetter CR, Noel D, Rubin B. Tobacco use prevalence and correlates among adolescents in a clinician initiated tobacco prevention trial in California, USA. J Epidemiol Community Health. 1996 Jun;50(3):340-6. doi: 10.1136/jech.50.3.340. PMID 8935468
- [Background] Hovell MF, Slymen DJ, Jones JA, Hofstetter CR, Burkham-Kreitner S, Conway TL, Rubin B, Noel D. An adolescent tobacco-use prevention trial in orthodontic offices. Am J Public Health. 1996 Dec;86(12):1760-6. doi: 10.2105/ajph.86.12.1760. PMID 9003134
- [Background] Wahlgren DR, Hovell MF, Slymen DJ, Conway TL, Hofstetter CR, Jones JA. Predictors of tobacco use initiation in adolescents: a two-year prospective study and theoretical discussion. Tob Control. 1997 Summer;6(2):95-103. doi: 10.1136/tc.6.2.95. PMID 9291217
- [Background] Hovell MF, Nichols JF, Irvin VL, Schmitz KE, Rock CL, Hofstetter CR, Keating K, Stark LJ. Parent/Child training to increase preteens' calcium, physical activity, and bone density: a controlled trial. Am J Health Promot. 2009 Nov-Dec;24(2):118-28. doi: 10.4278/ajhp.08021111. PMID 19928484
- [Background] Zakarian JM, Hovell MF, Conway TL, Hofstetter CR, Slymen DJ. Tobacco use and other risk behaviors: cross-sectional and predictive relationships for adolescent orthodontic patients. Nicotine Tob Res. 2000 May;2(2):179-86. doi: 10.1080/713688132. PMID 11072456
- [Background] Russos S, Hovell MF, Keating K, Jones JA, Burkham SM, Slymen DJ, Hofstetter CR, Rubin B. Clinician compliance with primary prevention of tobacco use: the impact of social contingencies. Prev Med. 1997 Jan-Feb;26(1):44-52. doi: 10.1006/pmed.1996.9994. PMID 9010897
- [Background] Slymen DJ, Hovell MF. Cluster versus individual randomization in adolescent tobacco and alcohol studies: illustrations for design decisions. Int J Epidemiol. 1997 Aug;26(4):765-71. doi: 10.1093/ije/26.4.765. PMID 9279608
- [Background] Hovell MF, Russos S, Beckhelm MK, Jones JA, Burkham-Kreitner SM, Slymen DJ, Hofstetter CR, Rubin B. Compliance with primary prevention in private practice: creating a tobacco-free environment. Am J Prev Med. 1995 Sep-Oct;11(5):288-93. PMID 8573357
- [Background] Russos S, Keating K, Hovell MF, Jones JA, Slymen DJ, Hofstetter CR, Rubin B, Morrison T. Counseling youth in tobacco-use prevention: determinants of clinician compliance. Prev Med. 1999 Jul;29(1):13-21. doi: 10.1006/pmed.1999.0495. PMID 10419794
- [Background] Hovell MF, Jones JA, Adams MA. The feasibility and efficacy of tobacco use prevention in orthodontics. J Dent Educ. 2001 Apr;65(4):348-53. PMID 11336120
- [Background] Morrison TC, Wahlgren DR, Hovell MF, Zakarian J, Burkham-Kreitner S, Hofstetter CR, Slymen DJ, Keating K, Russos S, Jones JA. Tracking and follow-up of 16,915 adolescents: minimizing attrition bias. Control Clin Trials. 1997 Oct;18(5):383-96. doi: 10.1016/s0197-2456(97)00025-1. PMID 9315423
- [Background] Keating KJ, Russos S, Hovell MF, Jones JA, Wahlgren D. Creating tobacco-free environments in clinicians' offices: Do patients notice? J Health Educ 2000;31(1):37-41.
- [Result] Cisse-Egbuonye N, Liles S, Schmitz KE, Kassem N, Irvin VL, Hovell MF. Availability of Vending Machines and School Stores in California Schools. J Sch Health. 2016 Jan;86(1):48-53. doi: 10.1111/josh.12349. PMID 26645420
- [Derived] Hovell MF, Schmitz KE, Liles S, Robusto K, Hofstetter CR, Nichols JF, Rock CL, Irvin V, Parker MS, Surillo SA, Noel D. A randomized controlled trial of orthodontist-based brief advice to prevent child obesity. Contemp Clin Trials. 2018 Jul;70:53-61. doi: 10.1016/j.cct.2018.05.003. Epub 2018 May 7. PMID 29747047